CLINICAL TRIAL: NCT03369548
Title: CirculAting Bile Acids as Biomarkers of Metabolic Health - Linking microbiotA, Diet and Health
Brief Title: CABALA Diet & Health Study
Acronym: CABALA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Reading (Other)
Collaborators: University College Cork (Other); Fondazione Edmund Mach (Other); Università degli Studi dell'Insubria (Other)
Responsible Party: Principal Investigator, Julie Lovegrove, Professor, University of Reading
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 17/47
Record Dates: First submitted 2017-12-01; First posted 2017-12-12 (Actual); Last update posted 2018-04-12 (Actual); Status verified 2018-04

CONDITIONS: Healthy
Keywords: Bile acids; Lipid metabolism; Cholesterol; Probiotics; Polyphenols; Prebiotics; Gut bacteria; Gut microbiota
MeSH Terms: interventions — Polyphenols; Prebiotics; Probiotics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Apple/ Polyphenol (Experimental): Participants will be asked to consume 2 Renetta Canada apples (with skin) and 2 placebo capsules every day for 8 weeks.
  Interventions: Other: Apple
- Oats / Prebiotic (Experimental): Participants will be asked to consume 40g jumbo rolled oats with semi-skimmed milk and 2 placebo capsules every day for 8 weeks.
  Interventions: Other: Oats
- Lactobacillus reuteri NCIMB 30242 / Probiotic (Experimental): Participants will be asked to consume 2 probiotic capsules and 40g cornflakes with semi-skimmed milk every day for 8 weeks.
  Interventions: Dietary Supplement: Lactobacillus reuteri NCIMB 30242
- Placebo / cornflakes (Placebo Comparator): Participants will be asked to consume 40g cornflakes with semi-skimmed milk and 2 placebo capsules every day for 8 weeks.
  Interventions: Other: Cornflakes

INTERVENTIONS:
Other: Apple — 2 Renetta Canada apples and 2 placebo capsules/ day
  Other Names: Polyphenol
  Arms: Apple/ Polyphenol
Other: Oats — 40g jumbo rolled oats with semi-skimmed milk and 2 placebo capsules / day
  Other Names: Prebiotic
  Arms: Oats / Prebiotic
Dietary Supplement: Lactobacillus reuteri NCIMB 30242 — 2 probiotic capsules and 40g cornflakes with semi-skimmed milk / day.
  Other Names: Probiotic
  Arms: Lactobacillus reuteri NCIMB 30242 / Probiotic
Other: Cornflakes — 40g cornflakes with semi-skimmed milk and 2 placebo capsules/ day.
  Other Names: Placebo
  Arms: Placebo / cornflakes

SUMMARY:
During digestion of fatty foods, the liver produces a substance called bile which helps with the absorption of fat in the gut (small intestine). Some research studies have shown that friendly bacteria that live in our gut can change the makeup of bile (referred to as bile acids) leading to a lowering of blood cholesterol levels, an important risk factor for developing heart disease. This finding has been found in people who consume diets high in dietary fibers and probiotics that enhance the growth of friendly gut bacteria, and also plant rich foods high in polyphenols (such as apples). At present, very little is known about how the makeup of bile acids can regulate blood cholesterol levels and if their measurement in blood, urine or stool samples can be used as an indicator of human health.

The aim of this study is to explore how consumption of foods which enhance the growth of friendly gut bacteria (such as probiotics, prebiotics, and plant rich foods high in polyphenols) can change the makeup of bile acids after 8 weeks. Changes in the bile acids measured in blood and stool samples will then be related to markers of health, such as blood cholesterol, glucose, insulin, vascular health and inflammatory markers.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* Aged 25-70 years
* BMI: 23-32 kg/m2
* Fasting glucose < 7 mmol/l
* Total cholesterol < 7.5 mmol/L
* Triglycerides < 2.3 mmol/L
* Habitual breakfast consumers
* Weight stable in the last three months

Exclusion Criteria:

* Smoker
* Diabetes
* Endocrine disease
* Cardiovascular disease diagnosis
* Gastrointestinal diseases
* Pancreatic, hepatic or renal diseases
* Medications that could influence study outcomes (e.g. lipid lowering medications, anti-depressants, anticoagulants)
* Antibiotic use within the last three months
* Food allergies (e.g. gluten, dairy, apples) and intolerances (e.g. lactose)
* Alcohol or drug abuse (Drink more than 14 units of alcohol per week)
* Anemia (men:haemoglobin<130g/ L and women <120 g/L
* Planning or currently on a weight reducing program
* Pregnancy, planned pregnancy in the next year or lactating
* Irregular menstrual cycle
* Planning or currently on a weight reducing program
* Currently taking part or participation in other research studies within the last three months
* Recent blood donation or unwilling to refrain from donating blood during the study
* Regular consumption of probiotic or prebiotic food supplements or fiber based laxatives and unwilling stop consuming these for the duration of the study

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2017-12-04 (Actual); Primary Completion 2019-11-30 (Estimated); Study Completion 2019-12-23 (Estimated)

PRIMARY OUTCOMES:
Circulating bile acids | Chronic and acute effects: Fasting and 6-hour postprandial response at both baseline and week 8
  Plasma bile acid profile

SECONDARY OUTCOMES:
Blood lipid profile | Chronic and acute effects: Fasting and 6-hour postprandial response at both baseline and week 8
  total, low density lipoprotein (LDL) and high density lipoprotein (HDL) cholesterol, triacylglycerol (TAG) and non-esterified fatty acids (NEFA)
Glucose response | Chronic and acute effects: Fasting and 6-hour postprandial response at both baseline and week 8
  Fasting and postprandial blood glucose concentrations
Insulin response | Chronic and acute effects: Fasting and 6-hour postprandial response at both baseline and week 8
  Fasting and postprandial blood insulin concentrations
C-peptide | Chronic and acute effects: Fasting and 6-hour postprandial response at both baseline and week 8
  Fasting and postprandial blood C-peptide concentrations
Inflammatory markers | Chronic and acute effects: Fasting and 6-hour postprandial response at both baseline and week 8
  Fasting blood concentrations of C-reactive protein (CRP), IL-18, IL-1β and tumour necrosis factor alpha (TNF-α)
Gut hormones | Chronic and acute effects: Fasting and 6-hour postprandial response at both baseline and week 8
  Fasting and postprandial concentrations of peptide YY, Glucagon-Like Peptide 1, Fibroblast growth factor 19
Metabolomics | Chronic and acute effects: Fasting and 6-hour postprandial response at both baseline and week 8
  Profile of metabolites in the blood (fasting and postprandial)
Nitric Oxide | Chronic and acute effects: Fasting and 6-hour postprandial response at both baseline and week 8
  Fasting and postprandial concentrations of nitric oxide
Cell-adhesion molecules | Chronic and acute effects: Fasting and 6-hour postprandial response at both baseline and week 8
  Fasting and postprandial concentrations of ICAM and VCAM
Short-chain fatty acids | Chronic and acute effects: Fasting and 6-hour postprandial response and faecal sample at both baseline and week 8
  Fasting and postprandial circulating short-chain fatty acids concentrations and fecal short-chain fatty acid concentrations
LDL receptor expression | This will be measured at baseline
  LDL receptor expression in peripheral blood mononuclear cells
Genotyping of bile acid receptor gene | This will be measured at baseline
  Genotyping of single-nucleotide polymorphisms (SNPs) in the FXR-encoding gene NR1H4
Platelets | Chronic and acute effects: Fasting and 6-hour postprandial response at both baseline and week 8
  Platelets will be collected for in-vitro studies
Gut microbiota | At baseline and week 8
  Next-generation sequencing of gut bacteria and enumeration of selected bacteria using FISH (fecal samples)
Bile acid excretion | At baseline and week 8
  Fecal bile acid concentrations
Energy excretion | At baseline and week 8
  Bomb calorimetry of fecal samples
Urine metabolites | At baseline and week 8
  Markers of intervention foods/ supplements in urine (24h urine collection)
Blood pressure and heart rate | Chronic and acute effects: Fasting and 6-hour postprandial response at both baseline and week 8
  Ambulatory blood pressure and heart rate
Body composition | At baseline and week 8
  Body composition measured using bio-impedance

CONTACTS AND LOCATIONS:
Overall Officials: Julie A Lovegrove, Professor, Principal Investigator — University of Reading
Locations (1):
- Hugh Sinclair Unit of Human Nutrition, Department of Food and Nutritional Sciences, University of Reading, Reading, Berkshire, United Kingdom

REFERENCES:
- [Derived] Alzoufairi S, Pushpass RG, Liu L, Lovegrove JA, Jackson KG. Impact of chronic consumption of probiotics, oats, and apples on expression of genes related to bile acids, lipid, gut peptides, and inflammation in peripheral monocular cells - findings from the CABALA study. Eur J Nutr. 2025 May 10;64(4):176. doi: 10.1007/s00394-025-03694-x. PMID 40347281